CLINICAL TRIAL: NCT07323849
Title: Tampa Scale for Kinesiophobia for Pelvic Pain (TSK-PP). Adaptation, Translation, and Psychometric Validation.
Brief Title: Tampa Scale for Kinesiophobia in Pelvic Pain (TSK-PP). Adaptation, Translation, and Psychometric Validation.
Status: Recruiting | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Borja Pérez-Domínguez, Associate Professor, University of Valencia
Other Study IDs: 2025-FIS-4201075
Record Dates: First submitted 2025-12-17; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Pelvic Pain
Keywords: Pelvic Pain; Kinesiophobia; Pain Measurement; Questionnaires / Psychometrics; Pain
MeSH Terms: conditions — Pelvic Pain; Kinesiophobia; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Pelvic Pain: Adults aged 18 years or older with chronic pelvic pain who are able to read and understand Spanish and have provided informed consent. This cohort will complete self-administered questionnaires to assess fear of movement (TSK-PP) and related psychometric measures.

SUMMARY:
The goal of this observational study is to adapt, translate, and evaluate the psychometric properties of the Tampa Scale for Kinesiophobia specifically for patients with pelvic pain (TSK-PP). The main questions it aims to answer are:

Can the TSK-PP reliably and validly measure fear of movement in individuals with pelvic pain?

Participants will complete standardized, self-administered questionnaires at a single point in time that assess:

Demographic and clinical characteristics (age, sex, marital status, medical diagnosis, duration and severity of pelvic pain) Fear of movement using the translated and adapted TSK-PP Fear-avoidance beliefs using the Fear-Avoidance Beliefs Questionnaire (FABQ) Pain catastrophizing using the Pain Catastrophizing Scale (PCS)

No interventions or treatments will be given as part of this study. The results will provide evidence on the reliability, validity, and clinical utility of the TSK-PP for use in research and practice with patients experiencing pelvic pain.

DETAILED DESCRIPTION:
Pelvic pain is a complex condition that can significantly impact daily functioning and quality of life. Fear of movement, or kinesiophobia, is recognized as a key psychological factor that may contribute to the transition from acute to chronic pain by promoting avoidance behaviors and limiting physical activity. Accurate measurement of kinesiophobia in patients with pelvic pain is essential for both clinical assessment and research purposes.

The Tampa Scale for Kinesiophobia (TSK) is a widely used instrument for assessing fear of movement, but its original items focus on general or musculoskeletal pain and do not capture the specific concerns of patients with pelvic pain. To address this gap, this study aims to adapt and translate the TSK for application in this population (TSK-PP) and evaluate its psychometric properties.

The study involves a rigorous process of cultural adaptation and translation, including item modification to reflect pelvic pain-specific contexts, forward translation into Spanish, independent review by an external expert, and back-translation into English to ensure conceptual equivalence. Following translation, the TSK-PP will be administered to adult patients with pelvic pain, alongside measures used for construct validation, including the Fear-Avoidance Beliefs Questionnaire (FABQ) and the Pain Catastrophizing Scale (PCS).

Data collected will include demographic and clinical characteristics such as age, sex, marital status, medical diagnosis, duration and severity of pelvic pain. These variables will allow for sample characterization and exploration of relationships with TSK-PP scores during psychometric evaluation.

This study will provide evidence on the reliability, validity, and applicability of the TSK-PP for assessing kinesiophobia in individuals with pelvic pain, supporting its use in both clinical practice and research settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Presence of chronic pelvic pain.
* Ability to read and understand Spanish.
* Signed informed consent provided prior to participation.

Exclusion Criteria:

* Inability to read or understand Spanish.
* Refusal or failure to provide informed consent for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from the adult population experiencing chronic pelvic pain. Eligible participants are adults aged 18 years or older who are able to read and understand Spanish and provide informed consent. The population includes individuals with varying demographic and clinical characteristics, such as age, sex, marital status, medical diagnosis, duration of pelvic pain, and pain severity. Participants will complete self-administered questionnaires at a single time point.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia | Baseline
  Fear of movement will be assessed using the Tampa Scale for Kinesiophobia adapted for patients with pelvic pain (TSK-PP), a translated and culturally adapted version of the original Tampa Scale for Kinesiophobia. The TSK-PP is a self-reported questionnaire consisting of 17 items, with total scores ranging from 17 to 68. Higher scores indicate greater levels of kinesiophobia (worse outcome).

SECONDARY OUTCOMES:
Fear-Avoidance Beliefs | Baseline
  Fear-avoidance beliefs will be assessed using the Fear-Avoidance Beliefs Questionnaire (FABQ), a self-reported instrument designed to evaluate beliefs about physical activity and work that may contribute to pain-related avoidance behaviors. The FABQ includes two subscales: Physical Activity (FABQ-PA; score range 0-24) and Work (FABQ-W; score range 0-42). Higher scores indicate stronger fear-avoidance beliefs (worse outcome).
Pain Catastrophizing | Baseline
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale (PCS), a self-reported questionnaire designed to measure catastrophic thinking related to pain, including rumination, magnification, and helplessness. The PCS total score ranges from 0 to 52, with higher scores indicating greater levels of pain catastrophizing (worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physiotherapy. University of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No